CLINICAL TRIAL: NCT07082829
Title: A Randomized, Double-blind, Sponsor-open, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Ascending Doses of ORX142 in Healthy Adults, Single Doses of ORX142 in Healthy Older Adults, and a Single Dose Crossover, Proof-of-concept Study of ORX142 in Acutely Sleep-deprived Healthy Subjects
Brief Title: A Study of ORX142 in Healthy Adult Subjects, Including Subjects 18 to 80 Years of Age
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centessa Pharmaceuticals (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORX142-0101
Record Dates: First submitted 2025-06-25; First posted 2025-07-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Excessive Daytime Sleepiness
Keywords: Excessive Daytime Sleepiness; orexin-2 receptor agonist
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (investigator- and subject-blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: SAD Study in Healthy Adults (Experimental)
  Interventions: Drug: ORX142 Tablets; Other: Placebo Tablets
- Part B: Food-effect Evaluation in Healthy Adults (Experimental)
  Interventions: Drug: ORX142 Tablets
- Part C: MAD Study in Healthy Adults (Experimental)
  Interventions: Drug: ORX142 Tablets; Other: Placebo Tablets
- Part D: Evaluation of a Single Dose in Healthy Older Adults (Experimental)
  Interventions: Drug: ORX142 Tablets; Other: Placebo Tablets
- Part E: PoC Study in Acutely Sleep-deprived Healthy Adults (Experimental)
  Interventions: Drug: ORX142 Tablets; Other: Placebo Tablets

INTERVENTIONS:
Drug: ORX142 Tablets — ORX142 Tablets
Other: Placebo Tablets — Placebo Tablets
  Arms: Part A: SAD Study in Healthy Adults; Part C: MAD Study in Healthy Adults; Part D: Evaluation of a Single Dose in Healthy Older Adults; Part E: PoC Study in Acutely Sleep-deprived Healthy Adults

SUMMARY:
Characterize the safety, tolerability and pharmacokinetics of ORX142 following single and multiple doses.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy males or females as determined by assessments at the Screening Visit.

   For Parts A, B, C, and E:

   a. Participants must be at least 18 years of age and no more than 55 years of age at the Screening
2. For Part D:

a .Participants must be at least 60 years of age and no more than 80 years of age at the Screening

Key Exclusion Criteria:

1. Presence of significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, malignancy, endocrine, neurological, or psychiatric disease, as determined by medical history, physical examination, and screening investigations.
2. History of seizure disorder, any other condition that increases the risk of seizure
3. Has a clinically significant sleep disorder, including insomnia or sleep apnea.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence and severity of Treatment-Emergent Adverse Events of oral single ascending doses of ORX142 in healthy adult subjects | From enrollment to the Follow-Up Visit 13 days post-discharge
  Safety and Tolerability as assessed by AEs and SAEs
Part B: Incidence and severity of Treatment-Emergent Adverse Events of oral single ascending doses of ORX142 in the fasted and fed states | From enrollment to the Follow-Up Visit 13 days post-discharge
  Safety and Tolerability as assessed by AEs and SAEs
Part C: Incidence and severity of Treatment-Emergent Adverse Events of oral multiple ascending doses of ORX142 in healthy adult subjects | From enrollment to the Follow-Up Visit 13 days post-discharge
  Safety and Tolerability as assessed by AEs and SAEs
Part D: Incidence and severity of Treatment-Emergent Adverse Events of oral single oral doses of ORX142 in healthy older adult subjects | From enrollment to the Follow-Up Visit 13 days post-discharge
  Safety and Tolerability as assessed by AEs and SAEs
Part E: Incidence and severity of Treatment-Emergent Adverse Events of oral of single oral doses of ORX142 in acutely sleep-deprived healthy adult subjects | From enrollment to the Follow-Up Visit 13 days post-discharge
  Safety and Tolerability as assessed by AEs and SAEs

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for ORX142 in subjects receiving ORX142 | Pre-dose and multiple post-dose timepoints, up to 48 hours
Tmax: Time of Maximum Concentration for ORX142 in subjects receiving ORX142 | Pre-dose and multiple post-dose timepoints, up to 48 hours
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for ORX142 in subjects receiving ORX142 | Pre-dose and multiple post-dose timepoints, up to 48 hours
T 1/2 (terminal elimination half-life): The time required for the terminal phase blood concentration of ORX142 to decrease by half in subjects receiving ORX142 | Pre-dose and multiple post-dose timepoints, up to 48 hours
Cmax: Maximum Observed Plasma Concentration for ORX142 in subjects receiving ORX142 in the fasted and fed state. | Pre-dose and multiple post-dose timepoints, up to 48 hours
Tmax: Time of Maximum Concentration for ORX142 in subjects receiving ORX142 in the fast and fed state | Pre-dose and multiple post-dose timepoints, up to 48 hours
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for ORX142 in subjects receiving ORX142 in the fast and fed state | Pre-dose and multiple post-dose timepoints, up to 48 hours
T 1/2 (terminal elimination half-life): The time required for the terminal phase blood concentration of ORX142 to decrease by half in subjects receiving ORX142 in the fast and fed state | Pre-dose and multiple post-dose timepoints, up to 48 hours
Mean sleep latency in the Maintenance of Wakefulness Test (MWT) for ORX142 versus placebo. | Part E: Day 2
Karolinska Sleepiness Scale score for ORX142 versus placebo | Part E: Day 1-2

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Site #1, Lincoln, Nebraska
  - Site #2, Eatontown, New Jersey
  - Site #3, New York, New York

IPD SHARING:
Plan to Share IPD: No